CLINICAL TRIAL: NCT05653947
Title: Cytokine Expression of IL-8 Before and After Root Canal Treatment in Patients With Symptomatic Apical Periodontitis: Clinical Trial
Brief Title: Expression of IL-8 Before and After Root Canal Treatment in Patients With Symptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Abouelenien, Lecturer of Endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: S.Abouelenien
Record Dates: First submitted 2022-11-27; First posted 2022-12-16 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Apical Periodontitis
Keywords: interleukin 8; apical periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vital teeth (Experimental): root canal instrumentation sodium hypochlorite 2.5% irrigation
  Interventions: Procedure: Root canal instrumentation, 2.5% NaOCl irrigation
- Non-vital teeth (Other): root canal instrumentation sodium hypochlorite 2.5% irrigation
  Interventions: Procedure: Root canal instrumentation, 2.5% NaOCl irrigation

INTERVENTIONS:
Procedure: Root canal instrumentation, 2.5% NaOCl irrigation — Root canal instrumentation, 2.5% NaOCl irrigation

SUMMARY:
This clinical study aimed to Compare the levels of Interleukin 8 before and after root canal treatment in patients with apical periodontitis

* Diagnosis
* Local anesthesia
* Isolation and disinfection of the tooth
* Two-staged access cavity preparation
* Patency of the root canals
* First sample collection using paper points
* Working length determination
* Chemico-mechanical preparation
* After 1 week, isolation, Second sample collection then obturation of the root canals and restoration of the tooth.
* Samples will be stored in (-80 C) freezer till collection of all samples then, quantification will be done using ELISA.

DETAILED DESCRIPTION:
Diagnosis:

* Personal data including name, address and phone number in addition to medical history and dental history will be collected from each patient in specific forms, then history of chief complaint will be recorded. The selected patients should show symptoms of symptomatic apical periodontitis (SAP) either associated with vital or necrotic teeth.
* Extra-oral and intra-oral clinical examination of the suspected tooth will be performed tentatively using a diagnostic mirror and probe.
* Radiograph will be taken using bisecting angle technique with a periapical digital sensor.
* The diagnosis of symptomatic apical periodontitis is confirmed through positive percussion test.
* After completing the diagnosis, the patient will be enrolled in the study.

Treatment procedure:

1. Local anesthesia: Anesthetizing the tooth using infiltration technique by local anesthesia (4% Articiane).
2. Isolation and disinfection: Operative field, including the tooth, the clamp, and rubber dam sheet will be disinfected using 30% hydrogen peroxide followed by 5% sodium hypochlorite solution. Subsequently, 5% sodium thiosulfate will be used to inactivate the disinfecting agents.
3. Access cavity preparation: a 2-stage access cavity preparation will be performed. The first stage involves the removal of caries and/or coronal restorations using sterile diamond bur. In the second stage, before entering the pulp chamber, the cavity will be disinfected according to the previous decontamination protocol. Then, a new round bur and tapered stone with round end will be used for access cavity preparation.

5. Patency of the root canal will be confirmed using stainless steel hand K-files size #10 and #15.

First sample collection: (PS-1) The pre-instrumentation periapical sample will be collected before cleaning and shaping by introducing a fine sterile size 15 paper point 2 mm beyond the canal terminus for 1 minute. This procedure will be performed twice. The paper points will be placed in a sterile micro-centrifugation tube, and immediately transferred to a -80 °C freezer until further testing.

6. Working length will be determined using an electronic apex locator then confirmed radiographically to be 1 mm shorter than radiographic apex. Then the canal will be enlarged to size #20.

7. Mechanical preparation will be performed using ProTaper Next rotary files in X-smart endodontic motor with adjusted speed (200rpm) and torque (2Ncm) according to the manufacturer's instructions.

The rotary files were introduced inside the canal using ethylenediaminetetraacetic acid (EDTA) gel with the following sequence:

* Orifice opener (size 40, taper 0.08) will be used to negotiate the coronal one-third of the canal is a slow downward movement without application of pressure.
* X1 (size 17, taper 0.04), will be used to negotiate the canal till the full working length is reached
* X2 (size 25, taper 0.06), will be used to full working length is reached
* X3 (size 30, taper 0.07), will be used to full working length is reached 8. The canal will be thoroughly irrigated with 2.5% sodium hypochlorite (NaOCl) root canal irrigant (5ml for 1 min) using disposable plastic syringe with side vented needle gauge 30 reaching 1 mm short of the working length. All teeth will receive the same volume of irrigant (5 ml prior to instrumentation, 5 ml between each file and 5 ml as final flush after root canal instrumentation to reach a total volume of 25 ml in total).

  9. The canal will then be dried by using sterile paper points and then flushed with 5 ml of saline to inactivate the NaOCl.

  10. The access cavity will be closed using sterile cotton pellet and temporary filling and patients will be recalled after 1 week.

  11. After 1 week, rubber dam will be applied Second sample collection: (PS-2) The post-instrumentation periapical sample will be collected following the same protocol mentioned. Then, master cone verification radiograph will be taken to ensure proper length and fit. Obturation will be done by modified single cone technique using epoxy resin sealer (Adseal) and 4% taper gutta percha cones together with auxillary cones.

  12. The access cavity will be restored with composite resin and occlusal contact will be checked.

  13. After collection of all the samples, quantification of IL-8 will be determined using ELISA kit before and after root canal instrumentation and irrigation. The kit is used according to the manufacturer's recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients
* Single canaled teeth diagnosed clinically with symptomatic apical periodontitis.
* Radiographic widening in the periodontal membrane space.
* Presence of pain on percussion.
* Patients' acceptance to participate in the trial.

Exclusion Criteria:

* Medically compromised patients.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively.
* Teeth that shows association with acute periapical abscess or swelling: Need special treatment steps which could involve additional visits with incision and drainage.
* Presence of periodontal disease
* Non restorability
* Immature teeth
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
interleukin 8 | immediately after access cavity preparation and immediately after root canal instrumentation
  Cytokine expression of IL8

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No